CLINICAL TRIAL: NCT02818309
Title: Efficacy and Safety of Lesogaberan (AZD3355) in Chinese Patients With Reflux Symptoms Refractory to Proton Pump Inhibitor Therapy: a Randomized Placebo-controlled Trial
Brief Title: Lesogaberan in Chinese Patients With Refractory Reflux Symptoms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201407100MIPA
Record Dates: First submitted 2016-06-21; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lesogaberan (Experimental): Lesogaberan
  Interventions: Drug: Lesogaberan
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lesogaberan — 120 mg bid
  Other Names: AZD3355
  Arms: Lesogaberan
Drug: Placebo — Placebo
  Other Names: Placebo for AZD3355
  Arms: Placebo

SUMMARY:
Lesogaberan may be used in Chinese GERD patients with partial response to PPI.

DETAILED DESCRIPTION:
To test the efficacy and safety of lesogaberan.

ELIGIBILITY:
Inclusion criteria

1. Provision of informed consent prior to any study specific procedures.
2. Male or female. Females of childbearing potential must have been using a highly effective contraceptive method for at least the previous 3 months.
3. Age 20-70 years, inclusive.
4. Body Mass Index (BMI) 18.5 - 35.0 kg/m2, inclusive.
5. Have at least 6 months history of Gastroesophageal reflux disease (GERD) symptoms (need not to have been consecutive) and endoscopy documented erosive esophagitis within 4 months.
6. Continuously treated during the last 8 weeks before enrolment with daily optimised unchanged standard dose proton pump inhibitor (PPI) therapy, such as esomeprazole 40 mg, lansoprazole 30 mg, dexlansoprazole 60 mg, rabeprazole 30 mg and pantoprazole 40 mg.
7. Able to read and write in the local language and use the e-diary device.
8. To be eligible for the screening phase the patients must have reported in the Reflux Symptom Questionnaire 7 day recall (RESQ-7) using 7 days recall of symptoms, a minimum of 3 days with a rating of at least moderate intensity on at least 1 of the following items; a burning feeling behind the breastbone or unpleasant movement of material upwards from the stomach.
9. To be eligible for randomisation the patients must have recorded in the Reflux Symptom Questionnaire electronic diary (RESQ-eD) on the last 7 days before randomisation, a minimum of 3 days with a symptom intensity of at least moderate on 1 of 2 items (a burning feeling behind the breastbone or an unpleasant movement of material upwards from the stomach), or any combination of both items (eg, 1 day on 1 item and 2 days on the other).

Exclusion criteria

1. Patients that had not experienced any GERD symptom improvement at all during PPI treatment.
2. Unstable or clinically significant cardiovascular (ischemic heart disease, congestive heart failure, arrhythmia), respiratory (chronic obstructive pulmonary disease), hepatic (AST or ALT or total bilirubin > upper limit of normal), renal (>1.5 mg/dL), metabolic (serum potassium or magnesium < lower reference range), psychiatric (major depression, schizophrenia) , or gastrointestinal and esophageal disorders besides GERD (peptic ulcer, eosinophilic esophagitis).
3. Current neurological disorders including nerve compression syndromes. Patients with well controlled migraine and other headache disorders could be included.
4. History of clinically significant orthostatic reaction or syncope.
5. History of a heart disease (including ischemic heart disease, congestive heart failure, cardiac arrhythmias, congenital long QT syndrome), or current signs or symptoms of any heart disease, or patients with clinically significant ECG abnormalities or QTcF >450 ms as determined by the investigator.
6. History of, or current malignant disease (radically treated basal cell cancer was allowed).
7. History of clinically significant electrolyte imbalances.
8. History of severe allergic or hypersensitivity reactions (such as Stevens Johnson syndrome, anaphylactic shock, angioedema-urticaria).
9. Using concomitant drugs that could potentially interfere with the pharmacodynamic effects of lesogaberan (such as baclofen or supplements containing GABA), alter gastrointestinal symptoms (such as type-2 histamine receptor agonists) or cause damage to the mucosal lining of the gastrointestinal tract (such as nonsteroidal anti-inflammatory drugs or acetylsalicylic acid >162 mg/day).
10. Prior surgery of the upper GI tract
11. Pregnant or breastfeeding females

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Treatment response as assessed by the symptom questionnaire RESQ-eD | 3 years
  Treatment response, defined as at most three days with heartburn or regurgitation of not more than mild intensity during the last 7 days of treatment based on RESQ-eD

SECONDARY OUTCOMES:
Time to treatment response as assessed by the symptom questionnaire RESQ-eD | 3 years
  time from the day of the first dose to the first of seven consecutive days meeting the responder definition
Time to sustained absence of symptoms as assessed by the symptom questionnaire RESQ-eD | 3 years
  time from the day of the first dose to the first of seven consecutive symptom-free days
The proportion of symptom-free days as assessed by the symptom questionnaire RESQ-eD | 3 years
The change from baseline for each separate symptom domain of the RESQ-eD | 3 years
Patients' consumption of rescue antacid medication over the 4 week treatment period | 3 years
Patient compliance with treatment determined by counts of returned unused capsules at each visit during the period of randomised treatment | 3 years
Subgroup analysis of in patients with different reflux profiles categorized by impedance-pH as assessed by the symptom questionnaire RESQ-eD | 3 years
  Treatment response, defined as at most three days with heartburn or regurgitation of not more than mild intensity during the last 7 days of treatment based on RESQ-eD
Number of participants with treatment-related adverse events as assessed by CRF_20150728 | 3 years
  Adverse events are any untoward medical occurrences in a patient or clinical trial subject to whom a medicinal product has been administered including occurrences which are not necessarily caused by or related to that product. According to previous studies, the common adverse events of lesogaberan include paraesthesia, diarrhea, pruritus, dizziness and nausea. The serious adverse events are defined as following: 1. results in death; 2.
  life-threatening; 3. requires hospitalisation or prolongation of existing hospitalisation; 4. results in persistent or significant disability or incapacity

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Huei Tseng, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will not open for public use.